CLINICAL TRIAL: NCT04480437
Title: Multi-parametric Breast Ultrasound Imaging as a Potential Biomarker for Breast Cancer
Acronym: mp-BUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-01-mp-BUS
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The proposed trial is designed as an explorative, open label, non-randomised, uncontrolled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Intervention (Experimental): mp-BUS data collection
  Interventions: Device: mp-BUS data collection

INTERVENTIONS:
Device: mp-BUS data collection — Collect ultrasound raw data and B-mode images of all kind of breast lesions to external storage device.

SUMMARY:
It is studied whether multi-parametric biomarkers such as speed-of-sound imaging or others, applied during breast ultrasound (BUS) imaging allows to classify lesions according to its malignancy. The standard reference intervention is BUS guided biopsy or the consensus of the board of experts judging the BUS imaging results if no biopsy is done.

DETAILED DESCRIPTION:
Patients with a palpable lump in the breast or suspicious findings in X-ray mammography typically undergo breast ultrasound examination as a supplemental imaging modality. Findings are then used for tumour classification according the American Collage of Radiology (ACR) Breast Imaging Reporting and Database System (BI-RADS) lexicon. Suspicious findings then undergo ultrasound-guided biopsy, which causes discomfort for the patient and introduces high emotional stress, and may involve - albeit very-small - risk of complications (such as bleeding and infections).

Today conventional breast ultrasound B-mode images do not have the specificity to reliably differentiate malignant and benign tissues in all cases and hence a biopsy intervention or close follow-up is necessitated. Multiparametric imaging bio-markers such as the novel method of speed-of-sound imaging may provide additional indicators to help to better classify lesions prior to biopsy and avoid any further work-up.

The study collects data with an ultrasound device during normal BUS examination which is then retrospectively processed to extract the desired multi-parametric BUS (mp-BUS) information of imaged tissue.

ELIGIBILITY:
Inclusion Criteria:

* Women who are suspected or suspected of having breast cancer and who are advised to perform a detailed breast ultrasound or tissue sampling (biopsy)
* Classification into groups:

  * Group 1: Foreseen for BUS guided biopsy
  * Group 2: BI-RADS classification I, II and III and foreseen for BUS only based diagnosis

Exclusion Criteria:

* Lactating women
* Women with mastitis
* Vulnerable persons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Speed-of-sound imaging shows malignancy of lesion | 6 months
  Evaluate the non-inferiority or superiority of the multi-parametric method compared to the standard ultrasound technique, using BUS guided biopsy as gold standard, to determine the malignancy of a lesion in woman breast.

CONTACTS AND LOCATIONS:
Overall Officials: Kubik Rahel, Prof. Dr., Principal Investigator — Kantonsspital Baden
Locations (1):
- Kantonsspital Baden, Baden, Switzerland

IPD SHARING:
Plan to Share IPD: No